CLINICAL TRIAL: NCT00000167
Title: Complications of Age-Related Macular Degeneration Prevention Trial (CAPT)
Brief Title: Complications of Age-Related Macular Degeneration Prevention Trial
Acronym: CAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Natalie Kurinij, NEI
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NEI-70
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-12

CONDITIONS: Macular Degeneration
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Laser treatment
  Interventions: Procedure: Low-Intensity Laser Treatment

INTERVENTIONS:
Procedure: Low-Intensity Laser Treatment — Initial: 60 barely visible burns, grid pattern. Re-treatment at 12 months: 30 barely visible burns, focal treatment.

SUMMARY:
To determine whether application of low-intensity laser treatment of eyes with drusen in the macula can prevent later complications of age-related macular degeneration and thereby preserve visual function.

DETAILED DESCRIPTION:
Complications of age-related macular degeneration (AMD) are the leading cause of severe vision loss among people aged 65 and over in the United States and many Western countries. Most, (approximately 90 percent), of this vision loss is due to the neovascular (or wet) form of AMD. The word neovascular describes the development of new, abnormal blood vessels in the back of the eye. Unfortunately, the majority of these new vessels are not amenable to currently available treatments.

The first sign that an eye may develop AMD is the presence of drusen, yellowish deposits under the retina. Current data suggests that eyes with large drusen are at increased risk for developing the vision threatening complications of AMD. Since the 1970s investigators have reported consistently that laser photocoagulation causes a reduction in large drusen. However, results of the effects of laser treatment on preventing later complications of AMD have been less consistent and based on relatively small numbers of patients.

Further study into the ability of a treatment to prevent vision loss from the advanced forms of AMD would have profound public health implications. A treatment that could reduce the risk of developing neovascularization by 30 percent might reduce the risk of blindness from AMD by one half. The Complications of Age-related Macular Degeneration Prevention Trial (CAPT) will assess whether treating drusen by laser photocoagulation reduces the risk of loss of visual acuity.

The CAPT is a multi-center, prospective, randomized clinical trial designed to assess the safety and effectiveness of low-intensity laser treatment in preventing vision loss among patients with large drusen in both eyes. A total of 1052 participants were enrolled in the study. Participants had one eye randomly assigned to laser treatment performed by a CAPT-certified ophthalmologist. The other eye was not treated. Both eyes were observed carefully for any changes for a period of five years. The effectiveness of the treatment was assessed using the following criteria:

Change in visual acuity (primary outcome measure of the study)

Incidence of complications of AMD such as neovascularization, serous detachment of the pigment epithelium, and geographic atrophy

Changes in contrast threshold and critical print size for reading

Quality of life assessments for patients, using the Visual Function Questionnaire 25 (VFQ-25), were conducted at the time of enrollment and at 5 years.

STUDY RESULTS:

Follow-up of patients was excellent; less than 3% of visual acuity examinations were missed. At 5 years, 188 (20.5%) treated eyes and 188 (20.5%) observed eyes had visual acuity scores ≥3 lines worse than at the initial visit (p= 1.00). The cumulative 5-year incidence rates for treated and observed eyes for CNV were 13.3% and 13.3% (p=0.95), respectively; and for GA were 7.4% and 7.8% (p=0.64), respectively. The contrast threshold doubled in 23.9% of treated eyes and in 20.5% of observed eyes (p=0.40). The critical print size doubled in 29.6% of treated eyes and in 28.4% of observed eyes (p=0.70). Seven (0.7%) treated eyes and 14 (1.3%) observed eyes had an adverse event of a ≥6 -line loss in visual acuity in the absence of late age-related macular degeneration or cataract.

As applied in CAPT, low intensity laser treatment did not demonstrate a clinically significant benefit on vision in eyes of people with bilateral large drusen.

ELIGIBILITY:
Patients eligible for CAPT can be either male or female and meet the following criteria:

Age at least 50 years old

Vision in each eye must measure 20/40 or better.

At least 10 large drusen in each eye

Available for follow-up examinations for 5 years after enrollment

Final eligibility is determined through a detailed eye examination by a CAPT-certified ophthalmologist.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 1999-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity (3-line loss) | 5 years

SECONDARY OUTCOMES:
Incidence of complications of AMD such as neovascularization, serous detachment of the pigment epithelium, and geographic atrophy | 5 years
Changes in contrast threshold and critical print size for reading | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Fine, MD, Study Chair — Scheie Eye Institute, The University of Pennsylvania School of Medicine
Locations (24):
- United States (24):
  - Retinal Consultants of Arizona, Ltd., Mesa, Arizona
  - Retinal Consultants of Arizona, Ltd., Peoria, Arizona
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - University of South Florida Eye Institute, Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Illinois Retina Associates, S.C., Harvey, Illinois
  - University of Iowa, Iowa City, Iowa
  - Ophthalmology & Visual Sciences at the University of Louisville, School of Medicine, Louisville, Kentucky
  - The Johns Hopkins University, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associate Retinal Consultants, P.C., Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - Retina-Vitreous Center, P.A., Edison, New Jersey
  - Retina-Vitreous Center, P.A., Lakewood, New Jersey
  - Southeast Clinical Research Associates, Charlotte, North Carolina
  - Retina Associates of Cleveland, Cleveland, Ohio
  - The Ohio State University, Department of Ophthalmology, Columbus, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Retina Northwest, P.C., Portland, Oregon
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Texas Retina Associates, Dallas, Texas
  - University of Wisconsin - Madison, Department of Ophthalmology and Visual Sciences, Madison, Wisconsin

REFERENCES:
- [Derived] Brader HS, Ying GS, Martin ER, Maguire MG; Complications of Age-Related Macular Degeneration Prevention Trial-CAPT Research Group. New grading criteria allow for earlier detection of geographic atrophy in clinical trials. Invest Ophthalmol Vis Sci. 2011 Nov 29;52(12):9218-25. doi: 10.1167/iovs.11-7493. PMID 22039251